CLINICAL TRIAL: NCT04487756
Title: Phase Ib/II Trial of the Combination of Atezolizumab With Dendritic Cell Vaccination as Maintenance Treatment in Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC) After Induction Treatment
Brief Title: Combination of Atezolizumab With Dendritic Cell Vaccine in Patients With Lung Cancer
Acronym: VENEZO-LUNG
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Oncológico Dr Rosell (Other)
Collaborators: Roche Pharma AG (Industry); Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOR-IISML42037; 2020-000448-72 (EudraCT Number)
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Small cell lung cancer; Atezolizumab; Dendritic cell vaccine; Safety; Efficacy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Injections; arginine decarboxylase; Vaccines; Carboplatin

STUDY DESIGN:
Intervention Model Description: single arm Phase Ib/II multicenter open label study, with translational sub-study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezo+DCvac (Experimental): - Induction (4 cycles, every 3 weeks): Carboplatin area under the curve (AUC) 5 (5 mg per milliliter per minute, administered intravenously on day 1 of each cycle) and etoposide (100 mg per square meter of body-surface area, administered intravenously on days 1 through 3 of each cycle) Atezolizumab, 1200 mg administered intravenously every 3 weeks on day 1 of each cycle)
  - Maintenance (only patients without PD after 4 induction cycles, up to PD): Atezolizumab iv (1200 mg/IV on day 1 every 3 weeks) DCV intradermally (max. 6 doses) on weeks 1, 3, 6, 9, 21, 33.
  Interventions: Drug: Atezolizumab 1200 mg in 20 ML Injection; Biological: ADC Vaccine; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab 1200 mg in 20 ML Injection — - Induction (4 cycles, every 3 weeks): Atezolizumab, 1200 mg administered intravenously every 3 weeks on day 1 of each cycle)
  - Maintenance (only patients without PD after 4 induction cycles, up to PD): Atezolizumab iv (1200 mg/IV on day 1 every 3 weeks)
  Other Names: Tecentriq
Biological: ADC Vaccine — - Maintenance (only patients without PD after 4 induction cycles, up to PD): DCV intradermally (max. 6 doses) on weeks 1, 3, 6, 9, 21, 33.
  Other Names: Autologous Dendritic cell (ADC) vaccine, Dendritic cell (DC) vaccine
Drug: Carboplatin — - Induction (4 cycles, every 3 weeks): Carboplatin AUC 5 (5 mg per milliliter per minute, administered intravenously on day 1 of each cycle) and etoposide (100 mg per square meter of body-surface area, administered intravenously on days 1 through 3 of each cycle)
  Other Names: Carboplatino (Teva/Accord/Pharmacia)

SUMMARY:
This is a single-arm Phase Ib/II multicenter open-label study, with translational sub-study, of atezolizumab plus autologous dendritic cell vaccine as maintenance treatment in extensive-stage small cell lung cancer (ES-SCLC). It is expected that three Spanish sites will include patients in this study.

Patients will receive standard treatment with carboplatin and etoposide, plus atezolizumab for four 21-day cycles (induction phase), followed by a maintenance phase during which they will receive the dendritic cell vaccine (6 doses maximum) in combination with atezolizumab until they had unacceptable toxic effects, disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, or no additional clinical benefit.

The two primary endpoints are the investigator-assessed toxicity and the 6 months PFS, both in the intention-to-treat population. Secondary Outcome Measures include: Duration of clinical benefit (DCB), Overall survival (OS) and Overall response rate (ORR)

The translational substudy will include:

Analysis of tumor tissue samples will consist of PD-L1 Immunohistochemistry testing, RNA expression, Work Environmental Scale (WES) analysis, and flow cytometry in pretreatment fresh tumor tissue.

The analysis will consist of T cell immunophenotyping, DC immunophenotyping, Tumoral RNA analysis by nanostring and tumoral cell-free DNA analysis by WES and cytokine analysis

DETAILED DESCRIPTION:
This is a single-arm Phase Ib/II multicenter open-label study, with translational sub-study, of atezolizumab plus autologous dendritic cell vaccine as maintenance treatment in extensive-stage small cell lung cancer (ES-SCLC). It is expected that three Spanish sites will include patients in this study.

Patients will receive standard treatment with carboplatin and etoposide, plus atezolizumab for four 21-day cycles (induction phase), followed by a maintenance phase during which they will receive atezolizumab and dendritic cell vaccine combination until they had unacceptable toxic effects, disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, or no additional clinical benefit. The two primary endpoints are the investigator-assessed toxicity and the 6 months PFS, both in the intention-to-treat population.

In the Phase Ib safety lead-in portion, up to 6 patients will be enrolled into and evaluated for dose-limiting toxicities (DLT) during the first 2 cycles of the maintenance therapy. If <2 out of 6 patients present with limiting toxicities, the administration of the investigational products will be deemed safe in the Phase 1b lead-in, therefore enrollment will be expanded into the Phase 2 cohort. Inclusion and treatment of up to 20 patients (including those enrolled in the Phase Ib lead-in) with atezolizumab and dendritic cell vaccination as maintenance therapy is finally expected.

Safety assessments will be based on adverse event reports, results of clinical laboratory tests, immune safety tests, physical examinations, vital sign measurements, Eastern Cooperative Oncology Group (ECOG) performance status both during the study, and up to six months following the last study drug administration. Adverse events (AEs) will be assessed throughout the study period and evaluated by using National Cancer Institute (NCI) Common Technology Criteria version of Adverse Events version 5.0 (NCI CTCAE v 5.0).

Tumor measurements will be performed by computed tomography (CT) scan at baseline, at week 6 (W6), at week 12 (W12), and every 9 weeks thereafter, to evaluate 6m PFS and response to treatment. The response will be evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) and the immune-related response criteria (irRECIST) as a secondary endpoint. Brain magnetic resonance imaging (MRI) will be performed at baseline (mandatory as per clinical practice), and along with CT scan at each timepoint, if there are brain metastasis at baseline.

Patients with stable disease (SD), partial response (PR) or complete response (CR) after induction with chemotherapy plus atezolizumab (CT scan on W12) will continue during the maintenance phase with atezolizumab plus dendritic cell vaccine.

Treatment with atezolizumab will continue until disease progression (PD), significant clinical deterioration, unacceptable toxicity, or if any criteria for withdrawal from the trial is fulfilled.

Treatment with dendritic cell vaccines will continue for a maximum of 6 doses until PD, significant clinical deterioration, unacceptable toxicity, or if any criteria for withdrawal from the trial are fulfilled (whichever occurs first).

Treatment may continue after the initial determination of PD per RECIST 1.1 if the subject's performance status remains stable, and if the opinion of the principal investigator, the subject will benefit from continued treatment and if other criteria are fulfilled as outlined in the protocol.

For patients who have a confirmed CR or PR, it should be considered prophylactic cranial irradiation (PCI) after completion of chemotherapy (i.e., induction) based on the investigator's judgment. Following the completion of the induction part, PCI may be administered concurrently with atezolizumab and dendritic cell vaccination during the maintenance part. For those patients who have not progressed at the time of study drug discontinuation, the tumor assessments (including all disease locations) will be assessed radiologically by CT or MRI, as performed at screening, every 9 weeks (approximately 63 ± 7 days), until the occurrence of PD or study completion. The same method of assessment (CT or MRI) should be used to characterize tumors at screening and at all follow-up assessments. If positron emission tomography (PET) is used, it should also be accompanied by spiral CT or MRI.

Safety will be defined based on the rate of serious adverse events (SAEs) comparing with historic controls of atezolizumab in monotherapy as a maintenance treatment.

Kaplan Meier method will be used to estimate the survival function. Translational study

Tumor samples: All patients will undergo baseline tumor tissue acquisition prior to enrollment. The only mandatory tissue biopsy is pretreatment. Tissue samples:

Pre induction treatment fresh and paraffin-embedded tumor sample (If obtaining a fresh biopsy is not feasible, the case should be discussed with Coordinating Investigators) Pre maintenance phase (for those that rebiopsy is feasible) After 24 weeks on maintenance phase (for those patents that continue on treatment after w24 on maintenance and rebiopsy is feasible) At tumor progression (for those patients who progressed and rebiopsy is feasible).

Analysis of tumor tissue samples will consist of PD-L1 Immunohistochemistry testing, RNA expression, WES analysis, and flow cytometry in pretreatment fresh tumor tissue.

Peripheral blood samples: Peripheral blood samples will be collected:

Pre induction treatment Pre maintenance phase After 9 weeks of the first vaccination At progression of the disease The analysis will consist of T cell immunophenotyping, DC immunophenotyping, Tumoral RNA analysis by nanostring and tumoral cell-free DNA analysis by WES and cytokine analysis

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of extensive-stage small cell lung cancer (ES-SCLC). Unequivocally confirmed diagnosis of SCLC by histology preferably including the presence of neuroendocrine features by immunohistochemistry.
2. Centrally confirmed tumor tissue viability for vaccine preparation.
3. No previous cancer treatment for advanced disease
4. Life expectancy at least 16 weeks
5. ECOG performance status 0 or 1.
6. Adequate normal organ and marrow function as defined below:

   Absolute neutrophil count ≥ 1.5 x 109 cells/L Platelets ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL Aspartate and alanine aminotransferases (AST, ALT) ≤ 2.5 x upper limit of normal (ULN) (≤ 5 x ULN, if documented liver metastases are present) Total bilirubin ≤ 2 x ULN (except patients with documented Gilbert's syndrome) Creatinine < 2 mg/dl (or a glomerular filtration rate > 60)
7. Prior palliative radiotherapy must have been completed at least 2 weeks prior to start the study treatment (subjects may receive localized palliative radiotherapy while receiving study drug).
8. Subjects with brain metastases are eligible if they are asymptomatic, are treated, or are neurological stable for at least 2 weeks without the use of steroids, or on a stable or decreasing dose of < 10 mg daily prednisone or equivalent.
9. Must be willing and able to accept one leukapheresis procedures
10. Written informed consent of approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the performance of any trial activities.
11. Male or female subjects aged ≥ 18 years.
12. Measurable disease by RECIST.1.1 criteria.
13. Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after the last atezolizumab treatment administration if the risk of conception exists.
14. Negative serum pregnancy test at screening for women of childbearing potential. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
15. Central negative serologic determination to HBsAg, Anti-HBc, HBV, HCV, HCV RNA, HIV-I RNA, Agp24 IIIV + AC IIIV ½ (MLIA) serum, IgG antigen core v. hepatitis B, RPR (Ac reaginic Lues-RPR, serum), Ac anti-HTLV I/II (if the patient came from an endemic zone), Ac anti-Trypanosoma Cruzi, Chagas, (if a patient came from the endemic zone), when RPR positive or doubtful for confirmation: IgG T. pallidum (ELISA) immunoglobulin M (IgM) T. pallidum (ELISA), when IgG T. Pallidum doubtful: Pt confirmatory immunoglobulin G (IgG)/IGM, T pallidum (LIA).

Exclusion Criteria:

1. Prior chemotherapy for extensive-stage ES-SCLC
2. Any prior anti-PD-1/PD-L1 antibody therapy
3. History of, or significant evidence of risk for, severe chronic inflammatory or autoimmune disease
4. Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed)
5. Human immunodeficiency virus (HIV) seropositivity, active Hepatitis B or C seropositivity
6. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
7. Pregnancy or breastfeeding; female patients must be surgically sterile or be postmenopausal for two years or must agree to use effective contraception during the period of treatment and 6 months after; all female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 24 hours from starting the conditioning chemotherapy; the definition of effective contraception will be based on the judgment of the study investigators; patients who are breastfeeding are not allowed on study
8. Any unresolved toxicity (CTCAE grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripheral neuropathy).
9. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. For phase I cohort, patients with autoimmune paraneoplastic syndromes will be also excluded.
10. Any syndrome that requires systemic corticosteroid/immunosuppressive medication EXCEPT for syndromes which would not be expected to recur in the absence of an external trigger (vitiligo, autoimmune thyroiditis, or type 1 diabetes mellitus are permitted to enroll)
11. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
12. History of primary immunodeficiency.
13. History of allogeneic organ transplant. 14 History of hypersensitivity to atezolizumab / ADC vaccine or any excipient.

15- Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diathesis including any subject known to have evidence of acute or chronic hepatitis B or C or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.

16- Known history of active tuberculosis. 17- Subjects with previous malignancies (except for non-melanoma skin cancer, and cancer in situ of the bladder, gastric, colon, cervical/dysplasia, melanoma, breast) are excluded unless a complete remission was achieved at least 5 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.

18- Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving atezolizumab.

19- Prior allogeneic stem-cell transplantation. 20- Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v 5.0), any history of anaphylaxis, or uncontrolled asthma.

21- Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of ADC + atezolizumab combination therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) rate at 6 months | At 6 months after start of treatment
  Calculated as the percentage of participants alive and without disease progression, as assessed by the Investigator using RECIST v1.1
Frequency and severity of AEs and SAEs (Safety) | Throughout the study. Approximately 3 years
  he number of patients with AEs and SAEs, changes in laboratory values, vital signs, ECGs, and results of physician examinations graded according to the CTCAE v 5.0.

SECONDARY OUTCOMES:
Duration of clinical benefit (DCB) as per RECIST 1.1 | Throughout the study. Approximately 3 years
  DCB calculated as the time (in months) from first dose of treatment to progression (or death from any cause) in patients who had a best overall response of CR, PR, or SD of ≥ 24 weeks.
Overall Survival (OS) | Throughout the study. Approximately 3 years
  Median Overall Survival (mOS) is calculated as the time from date of inclusion to date of death due to any cause.
Objective response rate (ORR1) as per RECIST 1.1 | Throughout the study. Approximately 3 years
  Rate of patients that achieve partial or complete response as best response during study induction treatment
Objective response rate (ORR2) as per RECIST 1.1 | Throughout the study. Approximately 3 years
  Rate of patients that have a further best response during maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: María González Cao, Study Chair — Hospital Quirón-Dexeus
Locations (3):
- Spain (3):
  - ICO Badalona, Badalona, Barcelona
  - Quirón Dexeus, Barcelona
  - Hospital Clínic Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No